



IRAS ID: 351150 - Chief Investigator: Dr Charles Prior

Participant Identification Number for this trial:

## **CONSENT FORM**

Title of Project: "Evaluation of spoken animation as a tool for imparting information about epidural labour analgesia" Name of Researcher: Dr Charles Prior

| | | | | | Please initial box |
|---|---|---|---|---|---|
| 1. | I confirm that I have read the information sheet dated (version 3) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | | |
| 3. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from the Queen Mary Maternity Unit, West Middlesex Hospital, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | | |
| 4. | I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. | | | | |
| 5. | I agree to my General Practitioner being informed of my participation in the study. / I agree to my General Practitioner being involved in the study, including any necessary exchange of information about me between my GP and the research team. | | | | |
| 6. | I understand that the information held and maintained by Chelsea & Westminster NHS Foundation Trust may be used to help contact me or provide information about my health status. | | | | |
| 7. | I agree to take part in the above study. | | | | |
| Name of Participant | | Date | <br>Si( | gnature | |
| Name of Researcher | | Date | <br>Sid | gnature | |